CLINICAL TRIAL: NCT00404872
Title: n-3 and Trans Fatty Acids and Major Cardiovascular Outcomes
Brief Title: Evaluating the Relationship Between Fatty Acids and Heart Disease
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Dariush Mozaffarian, MD, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 1363; R01HL085710 (NIH); R01HL085710-01 (NIH)
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Diseases; Heart Failure, Congestive; Atrial Fibrillation; Cerebrovascular Accident
Keywords: Stroke
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Atrial Fibrillation; Stroke

SUMMARY:
Cardiovascular disease (CVD) affects millions of people in the United States; each year, more people die from CVD than from any other disease. Individuals with low levels of n-3 fatty acids and high levels of trans-fatty acids may have an increased risk of developing CVD. This study will evaluate the link between fatty acids and the presence of CVD in older adults.

DETAILED DESCRIPTION:
CVD includes diseases that affect the heart and blood vessels, including congestive heart failure (CHF), atrial fibrillation (AF), and stroke. CVD may be associated with low levels of n-3 fatty acids and high levels of trans-fatty acids, but more research is needed to determine the role of various fatty acids in the development of CVD. Results from prior studies on this topic have not always been reliable because data from self-reported dietary questionnaires on fatty acid intake have sometimes been inaccurate. A more effective way to measure levels of fatty acids is to analyze blood samples. This study will use blood samples of participants in the Cardiovascular Health Study, a study that examined CVD risk factors in older adults, to determine the link between various fatty acids and the incidence of CHF, AF, and stroke. The results from this study may help researchers identify the dietary factors that influence the development of CVD in older adults.

This study will examine previously collected data from participants in the Cardiovascular Health Study. There will be no study visits specifically for this study. Plasma samples obtained from participants will be analyzed for the presence of n-3 fatty acids and trans-fatty acids. The study will also determine the incidence of CHF, AF, and stroke and the way in which fatty acids are related to hemodynamics, heart structure and function, electrophysiology, insulin sensitivity, inflammation, endothelial function, and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Cardiovascular Health Study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4766
Dates: Start 1989-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Mozaffarian, MD, DrPH, Principal Investigator — Harvard Medical School and Harvard School of Public Health
Locations (4):
- United States (4):
  - Channing Laboratory, Harvard Medical School, Boston, Massachusetts
  - Harvard School of Public Health, Boston, Massachusetts
  - Cardiovascular Health Research Unit, University of Washington, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Fried LP, Borhani NO, Enright P, Furberg CD, Gardin JM, Kronmal RA, Kuller LH, Manolio TA, Mittelmark MB, Newman A, et al. The Cardiovascular Health Study: design and rationale. Ann Epidemiol. 1991 Feb;1(3):263-76. doi: 10.1016/1047-2797(91)90005-w. PMID 1669507
- [Background] Tell GS, Fried LP, Hermanson B, Manolio TA, Newman AB, Borhani NO. Recruitment of adults 65 years and older as participants in the Cardiovascular Health Study. Ann Epidemiol. 1993 Jul;3(4):358-66. doi: 10.1016/1047-2797(93)90062-9. PMID 8275211